CLINICAL TRIAL: NCT01222247
Title: Antenatal Late Preterm Steroids (ALPS): A Randomized Placebo-Controlled Trial
Acronym: ALPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HL98354-HD36801-ALPS; U10HD021410 (NIH); U10HD027869 (NIH); U10HD027917 (NIH); U10HD053118 (NIH); U10HD027915 (NIH); U10HD034116 (NIH); U10HD034208 (NIH); U10HD053097 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U10HD036801 (NIH); U01HL098354 (NIH); U01HL098554 (NIH); U10HD068268 (NIH); U10HD068258 (NIH); U10HD068282 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy; Respiratory Distress Syndrome; Pregnancy Outcomes; Preterm Birth
Keywords: Betamethasone; Steroids; Perinatology; Late Preterm
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — Betamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Betamethasone (Active Comparator): A course of two 2mL intramuscular (IM) injections containing 3 mg of betamethasone, 24 hours apart
  Interventions: Drug: Betamethasone
- Placebo (Placebo Comparator): A similar course of an identical appearing placebo: two 2 mL IM injections of placebo, 24 hours apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Betamethasone — The active study drug, betamethasone. 3 mg per ml betamethasone sodium phosphate 3 mg per milliliter betamethasone acetate The first dose of study drug medication will be administered at randomization as 2 ml injection; the next dose of 2 ml will be administered 24 hours later.
  Other Names: Corticosteroid
  Arms: Betamethasone
Drug: Placebo — Similar course of identical appearing placebo: 2 mL IM injections, 24 hours apart.
  Arms: Placebo

SUMMARY:
This is a randomized placebo controlled trial to evaluate whether antenatal corticosteroids can decrease the rate of neonatal respiratory support, thus decreasing the rate of NICU admissions and improving short-term outcomes in the late preterm infant. The use of antenatal corticosteroids has been shown to be beneficial in women at risk for preterm delivery prior to 34 weeks but has not been evaluated in those likely to deliver in the late preterm period

DETAILED DESCRIPTION:
The rate of preterm birth has steadily increased in the United States over the past 10 years. This increase is driven in part by the rising rate of late preterm birth, defined as those births occurring between 34 and 36 weeks. Late preterm infants experience a higher rate of readmission than their term counterparts, and these infants are more likely to suffer complications such as respiratory distress, kernicterus, feeding difficulties, and hypoglycemia. Late preterm infants also have a higher mortality for all causes when compared to term infants. The use of antenatal corticosteroids has been shown to be beneficial in women at risk for preterm delivery prior to 34 weeks but has not been evaluated in those likely to deliver in the late preterm period. If shown to reduce the need for respiratory support and thus to decrease the rate of special care nursery admissions and improve short-term outcomes, the public health and economic impact will be considerate.This protocol describes a randomized placebo controlled trial to evaluate whether antenatal corticosteroids can decrease the rate of neonatal respiratory support, thus decreasing the rate of neonatal intensive care unit (NICU) admissions and improving short-term outcomes in the late preterm infant.

Two follow-up studies will be conducted concurrently. The first follow-up study will examine if the positive effects of betamethasone on lung function will persist in children at 6 years of age of mothers randomized to betamethasone with an expected late preterm delivery. Neonatal respiratory morbidity is associated with an increased risk of adverse childhood respiratory disease. Thus it is quite plausible that the effect of betamethasone, in reducing neonatal morbidity, particularly TTN, will translate into improved respiratory morbidity in early childhood.The primary outcome is childhood respiratory disease defined by a composite outcome of abnormal pulmonary function test (PFT) measured by spirometry, physician diagnosis of asthma, or other respiratory illnesses with medication.

The second follow-up study will examine whether late preterm antenatal betamethasone treatment is associated with long-term neurocognitive functioning, and whether there are any long-term consequences of what is believed to be transient neonatal hypoglycemia. Cognitive function will be measured by the Differential Ability Scales 2nd Edition (DAS-II) core components of the general conceptual ability (GCA) that includes verbal ability, non-verbal reasoning ability and spatial ability. The primary outcome is defined as a GCA score of <85 (1 standard deviation below the mean) at 6 years of age or greater.

ELIGIBILITY:
Inclusion Criteria:

Singleton Pregnancy. A twin pregnancy reduced to singleton (either spontaneously or therapeutically) before 14,0 weeks by project gestational age is acceptable

Gestational age at randomization between 34,0 weeks and 36,5 weeks confirmed by study criteria

High probability of delivery in the late preterm period (any one of the following):

* Membrane rupture as defined by the occurrence of any two of the following: pooling of fluid in the vaginal vault, positive Nitrazine test, ferning of vaginal fluid, positive AmniSure test; or any one of the following: indigo carmine pooling in the vagina after amnioinfustion, visible leakage of amniotic fluid from the cervix

or

* Preterm labor with intact membranes. Preterm labor is defined as at least 6 regular uterine contractions in an observation period of no more than 60 minutes and at least one of the following: cervix greater than or equal to 3cm dilated or at least 75% effaced

or

* Planned delivery by induction of labor or cesarean section in no less than 24 hours and no more than 7 days, as deemed necessary by the provider. An induction must be scheduled to start by 36,5 weeks at the latest, whereas a cesarean delivery must be scheduled by 36,6 weeks at the latest. Therefore the latest gestational age for randomization is 36,4 weeks for a planned induction. The planned delivery may be for any indication, such as the following: prior myomectomy, prior classical cesarean, intrauterine growth restriction (IUGR), oligohydramnios, preeclampsia, nonreassuring fetal heart rate tracing warranting delivery, abruption, placenta previa

Exclusion Criteria:

1. Any prior antenatal corticosteroid course during the pregnancy because of potential contamination of the placebo group
2. Candidate for stress dose corticosteroids because of chronic steroid therapy to prevent suppression of adrenal gland, because of potential contamination of the placebo group
3. Twin gestation reduced to a singleton gestation at or after 14 weeks 0 days by project gestational age either spontaneously or therapeutically
4. Fetal demise, or known major fetal anomaly, including cardiac anomaly and hydrops
5. Maternal contraindication to betamethasone: hypersensitivity reaction to any components of the medication, idiopathic thromboycytopenic purpura, systemal fungal infection in case of exacerbation by betamethasone, use of amphotericin B due to the possibility of heart failure with concomitant betamethasone
6. Pre-gestational diabetes - exclude if the patient was on medication (insulin, glyburide) prior to pregnancy
7. Delivery expected within 12 hours of randomization, because of insufficient time of corticosteroids to confer benefit, including any of the following:

   A. Rupture of Membranes (ROM) does not satisfy protocol criteria - exclude if the patient being evaluated for Preterm Premature Rupture of Membranes (pPROM), does not have preterm labor or planned delivery and does not satisfy the spontaneous membrane rupture criteria (any 2 of: positive Nitrazine test, pooling of fluid in the vaginal vault test or ferning of vaginal fluid; or indigo carmine pooling in the vagina after amnioinfusion; or visible leakage of amniotic fluid from the cervix) B. Rupture of the membranes in the presence of more than 6 contractions per hour or cervical dilation of 3 cm or more, unless oxytocin was withheld for at least 12 hours (other induction agents allowed) C. Chorioamnionitis - exclude if patient is diagnosed with chorioamnionitis D. Cervical dilation ≥ 8 cm E. Evidence of non-reassuring fetal status requiring immediate delivery
8. Participation in another interventional study that influences neonatal morbidity and mortality
9. Participation in this trial in a previous pregnancy
10. Delivery at a non-network hospital
11. At 36, 0 weeks to 36, 5 weeks and quota for 36 weeks already met. To ensure there is an adequate proportion of women presenting at 34 to 35 weeks of gestation, enrollment will be restricted so that no more than 50% of the women in the trial present at 36 weeks.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2831 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Longo, MD, Study Director — NICHD Project Scientist; Rebecca Clifton, PhD, Principal Investigator — George Washington University; Cynthia Gyamfi Bannerman, MD, Study Chair — Columbia University
Locations (17):
- United States (17):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Wayne State University, Detroit, Michigan
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas - Southwest, Dallas, Texas
  - University of Texas - Galveston, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after completion and publication of the main analyses per NIH policy. Requests can be sent to mfmudatasets@bsc.gwu.edu.

REFERENCES:
- [Background] Davidoff MJ, Dias T, Damus K, Russell R, Bettegowda VR, Dolan S, Schwarz RH, Green NS, Petrini J. Changes in the gestational age distribution among U.S. singleton births: impact on rates of late preterm birth, 1992 to 2002. Semin Perinatol. 2006 Feb;30(1):8-15. doi: 10.1053/j.semperi.2006.01.009. PMID 16549207
- [Background] Raju TN, Higgins RD, Stark AR, Leveno KJ. Optimizing care and outcome for late-preterm (near-term) infants: a summary of the workshop sponsored by the National Institute of Child Health and Human Development. Pediatrics. 2006 Sep;118(3):1207-14. doi: 10.1542/peds.2006-0018. PMID 16951017
- [Background] Escobar GJ, Clark RH, Greene JD. Short-term outcomes of infants born at 35 and 36 weeks gestation: we need to ask more questions. Semin Perinatol. 2006 Feb;30(1):28-33. doi: 10.1053/j.semperi.2006.01.005. PMID 16549211
- [Background] Hamilton BE, Ventura SJ, Martin JA, and Sutton PD. Preliminary births for 2004. Health E-stats. Hyattsville, MD: National Center for Health Statistics. Released October 28, 2005.
- [Background] Buus-Frank ME. The great imposter. Adv Neonatal Care. 2005 Oct;5(5):233-6. doi: 10.1016/j.adnc.2005.08.012. No abstract available. PMID 16202965
- [Background] Hoyert DL, Mathews TJ, Menacker F, Strobino DM, Guyer B. Annual summary of vital statistics: 2004. Pediatrics. 2006 Jan;117(1):168-83. doi: 10.1542/peds.2005-2587. PMID 16396875
- [Background] Dudell GG, Jain L. Hypoxic respiratory failure in the late preterm infant. Clin Perinatol. 2006 Dec;33(4):803-30; abstract viii-ix. doi: 10.1016/j.clp.2006.09.006. PMID 17148006
- [Background] Laptook A, Jackson GL. Cold stress and hypoglycemia in the late preterm ("near-term") infant: impact on nursery of admission. Semin Perinatol. 2006 Feb;30(1):24-7. doi: 10.1053/j.semperi.2006.01.014. PMID 16549210
- [Background] Neu J. Gastrointestinal maturation and feeding. Semin Perinatol. 2006 Apr;30(2):77-80. doi: 10.1053/j.semperi.2006.02.007. PMID 16731281
- [Background] Bhutani VK, Johnson L. Kernicterus in late preterm infants cared for as term healthy infants. Semin Perinatol. 2006 Apr;30(2):89-97. doi: 10.1053/j.semperi.2006.04.001. PMID 16731283
- [Background] Moster D, Lie RT, Markestad T. Long-term medical and social consequences of preterm birth. N Engl J Med. 2008 Jul 17;359(3):262-73. doi: 10.1056/NEJMoa0706475. PMID 18635431
- [Background] McIntire DD, Leveno KJ. Neonatal mortality and morbidity rates in late preterm births compared with births at term. Obstet Gynecol. 2008 Jan;111(1):35-41. doi: 10.1097/01.AOG.0000297311.33046.73. PMID 18165390
- [Background] Kramer MS, Demissie K, Yang H, Platt RW, Sauve R, Liston R. The contribution of mild and moderate preterm birth to infant mortality. Fetal and Infant Health Study Group of the Canadian Perinatal Surveillance System. JAMA. 2000 Aug 16;284(7):843-9. doi: 10.1001/jama.284.7.843. PMID 10938173
- [Background] Gray RF, Indurkhya A, McCormick MC. Prevalence, stability, and predictors of clinically significant behavior problems in low birth weight children at 3, 5, and 8 years of age. Pediatrics. 2004 Sep;114(3):736-43. doi: 10.1542/peds.2003-1150-L. PMID 15342847
- [Background] Linnet KM, Wisborg K, Agerbo E, Secher NJ, Thomsen PH, Henriksen TB. Gestational age, birth weight, and the risk of hyperkinetic disorder. Arch Dis Child. 2006 Aug;91(8):655-60. doi: 10.1136/adc.2005.088872. Epub 2006 Jun 5. PMID 16754656
- [Background] Clark RH. The epidemiology of respiratory failure in neonates born at an estimated gestational age of 34 weeks or more. J Perinatol. 2005 Apr;25(4):251-7. doi: 10.1038/sj.jp.7211242. PMID 15605071
- [Background] Stutchfield P, Whitaker R, Russell I; Antenatal Steroids for Term Elective Caesarean Section (ASTECS) Research Team. Antenatal betamethasone and incidence of neonatal respiratory distress after elective caesarean section: pragmatic randomised trial. BMJ. 2005 Sep 24;331(7518):662. doi: 10.1136/bmj.38547.416493.06. Epub 2005 Aug 22. PMID 16115831
- [Background] Rubaltelli FF, Dani C, Reali MF, Bertini G, Wiechmann L, Tangucci M, Spagnolo A. Acute neonatal respiratory distress in Italy: a one-year prospective study. Italian Group of Neonatal Pneumology. Acta Paediatr. 1998 Dec;87(12):1261-8. doi: 10.1080/080352598750030951. PMID 9894827
- [Background] Yoder BA, Gordon MC, Barth WH Jr. Late-preterm birth: does the changing obstetric paradigm alter the epidemiology of respiratory complications? Obstet Gynecol. 2008 Apr;111(4):814-22. doi: 10.1097/AOG.0b013e31816499f4. PMID 18378739
- [Background] Tita AT, Landon MB, Spong CY, Lai Y, Leveno KJ, Varner MW, Moawad AH, Caritis SN, Meis PJ, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai BM, Langer O, Thorp JM, Ramin SM, Mercer BM; Eunice Kennedy Shriver NICHD Maternal-Fetal Medicine Units Network. Timing of elective repeat cesarean delivery at term and neonatal outcomes. N Engl J Med. 2009 Jan 8;360(2):111-20. doi: 10.1056/NEJMoa0803267. PMID 19129525
- [Background] Wang ML, Dorer DJ, Fleming MP, Catlin EA. Clinical outcomes of near-term infants. Pediatrics. 2004 Aug;114(2):372-6. doi: 10.1542/peds.114.2.372. PMID 15286219
- [Background] Shapiro-Mendoza CK, Tomashek KM, Kotelchuck M, Barfield W, Weiss J, Evans S. Risk factors for neonatal morbidity and mortality among "healthy," late preterm newborns. Semin Perinatol. 2006 Apr;30(2):54-60. doi: 10.1053/j.semperi.2006.02.002. PMID 16731277
- [Background] Tomashek KM, Shapiro-Mendoza CK, Weiss J, Kotelchuck M, Barfield W, Evans S, Naninni A, Declercq E. Early discharge among late preterm and term newborns and risk of neonatal morbidity. Semin Perinatol. 2006 Apr;30(2):61-8. doi: 10.1053/j.semperi.2006.02.003. PMID 16731278
- [Result] Gyamfi-Bannerman C, Thom EA, Blackwell SC, Tita AT, Reddy UM, Saade GR, Rouse DJ, McKenna DS, Clark EA, Thorp JM Jr, Chien EK, Peaceman AM, Gibbs RS, Swamy GK, Norton ME, Casey BM, Caritis SN, Tolosa JE, Sorokin Y, VanDorsten JP, Jain L; NICHD Maternal-Fetal Medicine Units Network. Antenatal Betamethasone for Women at Risk for Late Preterm Delivery. N Engl J Med. 2016 Apr 7;374(14):1311-20. doi: 10.1056/NEJMoa1516783. Epub 2016 Feb 4. PMID 26842679
- [Derived] Laptook AR, Chalak L, Pappas A, Davis A, Sanchez PJ, Van Meurs KP, Oh W, Sommers R, Shankaran S, Hensman AM, Rouse DJ, McDonald S, Das A, Goldberg RN, Ambalavanan N, Gyamfi-Bannerman C, Thom EA, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network (NRN); Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units (MFMU) Network. The effects of betamethasone on the amplitude integrated EEG of infants born at 34- or 35-weeks gestation. J Perinatol. 2022 Dec;42(12):1615-1621. doi: 10.1038/s41372-022-01415-4. Epub 2022 May 26. PMID 35618748
- [Derived] McGoldrick E, Stewart F, Parker R, Dalziel SR. Antenatal corticosteroids for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2020 Dec 25;12(12):CD004454. doi: 10.1002/14651858.CD004454.pub4. PMID 33368142
- See also: (The public website of the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal Fetal Medicine Units (MFMU) Network) — http://www.bsc.gwu.edu/mfmu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from October 2010 to February 2015 at 17 university-based clinical centers. Women with a singleton pregnancy at 34 weeks 0 days to 36 weeks 5 days of gestation and a high probability of delivery in the late preterm period were eligible to be enrolled.
Period: Overall Study
Arm/Group | Betamethasone | Placebo
Started | 1429 | 1402
Received 2 Doses | 860 | 826
Received 1 Dose | 568 | 571
Did Not Receive Assigned Medication | 1 | 5
Completed | 1427 | 1400
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Betamethasone | Placebo | Total
Number analyzed (Participants) | 1429 | 1402 | 2831
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean maternal age | 28.6 (6.3) | 27.8 (6.1) | 28.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1429 | 1402 | 2831
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 376 | 381 | 757
  White | 828 | 800 | 1628
  Hispanic | 168 | 182 | 350
  Other, unknown, more than one race | 57 | 39 | 96
Region of Enrollment [Number; unit: participants]
  United States | 1429 | 1402 | 2831
Indication for trial entry [Count of Participants; unit: Participants]
  Preterm labor with intact membranes | 400 | 392 | 792
  Ruptured membranes | 316 | 304 | 620
  Exp delivery for gestational HTN or preeclampsia | 370 | 385 | 755
  Expected delivery for fetal growth restriction | 46 | 48 | 94
  Expected delivery for oligohydramnios | 50 | 42 | 92
  Expected delivery for other indication | 247 | 231 | 478
Gestational age at trial entry [Count of Participants; unit: Participants]
  ≤34 weeks 6 days | 369 | 399 | 768
  35 weeks 0 days to 35 weeks 6 days | 571 | 532 | 1103
  ≥36 weeks 0 days | 489 | 471 | 960
Smoking during pregnancy [Count of Participants; unit: Participants] | 204 | 186 | 390
Nulliparous [Count of Participants; unit: Participants] | 457 | 448 | 905
Preeclampsia or gestational hypertension [Count of Participants; unit: Participants] | 433 | 440 | 873
Gestational diabetes [Count of Participants; unit: Participants] | 153 | 153 | 306
Major congenital anomaly in infant [Count of Participants; unit: Participants] — Although the presence of a major congenital anomaly was an exclusion criterion, these disorders were not discovered until birth. Therefore we report this as a baseline measure on the publication and not an outcome. To be consistent with the publication, we report this as a baseline measure here.
  Participants | 11 | 21 | 32

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Composite Outcome
Description: Need for respiratory support: Continuous positive airway pressure (CPAP) or humidified high-flow nasal cannula (HHFNC) for greater than or equal to 2 hours or more in the first 72 hours, or fraction of inspired oxygen (FiO2) greater than or equal to 0.30 for 4 hours or more in the first 72 hours, or mechanical ventilation in the first 72 hours, or Extracorporeal membrane oxygenation (ECMO) Stillbirth, or neonatal death less than 72 hours of age
Time Frame: 72 hours of life
Population: The number of participants analyzed accounts for the 4 participants for which baseline measures were obtained but who were subsequently lost to follow-up (2 in each group).
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants
  Primary Outcome Composite | 165 | 202
  CPAP or high-flow cannula ≥2 continuous hrs | 145 | 184
  Fraction of inspired O2 of ≥0.30 for ≥4 cont hrs | 48 | 61
  Mechanical ventilation | 34 | 43
  Extracorporeal membrane oxygenation (ECMO) | 0 | 0
  Stillbirth or neonatal death ≤72 hr after birth | 0 | 0
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Analysis for Primary Outcome composite; Test type: Superiority or Other; p = 0.02, Chi-squared; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.66 to 0.97]
Statistical Analysis 2: Comparison: Betamethasone vs Placebo; Analysis for CPAP or high-flow nasal cannula; Test type: Superiority; p = 0.01, Chi-squared; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.63 to 0.95]
Statistical Analysis 3: Comparison: Betamethasone vs Placebo; Analysis for Fraction of inspired oxygen; Test type: Superiority; p = 0.17, Chi-squared; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.53 to 1.12]
Statistical Analysis 4: Comparison: Betamethasone vs Placebo; Analysis for mechanical ventilation; Test type: Superiority; p = 0.26, Chi-squared; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.50 to 1.21]

2. Secondary Outcome: Number of Neonates With Severe Respiratory Complication,
Description: A severe respiratory complication was defined as any of the following occurrences within 72 hours after birth: CPAP or high-flow nasal cannula for at least 12 hours, supplemental oxygen with a fraction of inspired oxygen of 0.30 or more for at least 24 hours, mechanical ventilation, stillbirth or neonatal death, or the need for ECMO. Except for the duration of CPAP or high-flow nasal cannula and the duration of a fraction of inspired oxygen of 0.30 or more, the criteria for a severe respiratory complication overlap with those of the primary outcome.
Time Frame: 72 hours of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants
  Severe Respiratory Complication Composite | 114 | 169
  CPAP or high-flow cannula ≥12 continuous hrs | 93 | 147
  Fraction of inspired 02 of ≥0.30 for ≥24 cont hrs | 20 | 34
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.53 to 0.84]

3. Secondary Outcome: Neonates Needing Immediate Resuscitation After Birth
Description: Need for resuscitation after birth: any intervention in the first 30 minutes other than blow-by oxygen
Time Frame: Within the first 30 minutes of birth
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1422 | 1390
Participants | 206 | 260
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.003, Chi-squared; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.66 to 0.92]

4. Secondary Outcome: Number of Neonates With Respiratory Distress Syndrome
Description: Respiratory distress defined as the presence of clinical signs of respiratory distress (tachypnea, retractions, flaring, grunting, or cyanosis) with an oxygen requirement and a chest x-ray that shows hypoaeration and reticulogranular infiltrates
Time Frame: Delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 79 | 89
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.36, Chi-squared; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.65 to 1.17]

5. Secondary Outcome: Number of Neonates With Transient Tachypnea of the Newborn
Description: TTN is defined as signs of respiratory distress, specifically tachypnea, that are resolved by 72 hours of age. TTN may be diagnosed in the absence of a chest X-ray or with a chest X-ray that is normal or shows signs of increased perihilar interstitial markings
Time Frame: by 72 hours after delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 95 | 138
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.002, Chi-squared; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.53 to 0.87]

6. Secondary Outcome: Number of Infants With Neonatal Apnea
Description: Neonatal apnea with respiratory pauses of more than 20 seconds duration resulting in bradycardia or oxygen desaturation below baseline.
Time Frame: 72 hours of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 33 | 37
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.57, Chi-squared; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.55 to 1.39]

7. Secondary Outcome: Number of Infants withChronic Lung Disease / Bronchopulmonary Dysplasia (BPD) Requiring Supplemental Oxygen
Description: Infants requiring supplemental oxygen of more than 0.21 for the first 28 days of life
Time Frame: 28 days of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 2 | 9
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.04, Chi-squared; Risk Ratio (RR) = 0.22, 95% CI 2-sided [0.02 to 0.92]

8. Secondary Outcome: Neonates With Pneumonia
Description: Neonatal pneumonia
Time Frame: by 72 hours of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 6 | 13
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.10, Chi-squared; Risk Ratio (RR) = 0.45, 95% CI 2-sided [0.17 to 1.19]

9. Secondary Outcome: Number of Neonates Needing Surfactant Administration
Description: Administration of surfactant for neonatal respiratory treatment
Time Frame: Delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 26 | 43
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.03, Chi-squared; Risk Ratio (RR) = 0.59, 95% CI 2-sided [0.37 to 0.96]

10. Secondary Outcome: Neonatal Outcome Composite
Description: Transient tachypnea of the newborn (TTN), respiratory distress syndrome (RDS), and apnea
Time Frame: 72 hours of life
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 198 | 249
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.004, Chi-squared; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.66 to 0.93]

11. Secondary Outcome: Number of Neonates With Pulmonary Air Leak
Description: Neonatal pulmonary air leak syndrome
Time Frame: 72 hours post delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 5 | 6
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.74, Chi-squared; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.25 to 2.68]

12. Secondary Outcome: Neonatal Death After 72 Hours of Delivery
Description: Neonatal death after 72 hours of life but before hospital discharge.
Time Frame: 72 hours after delivery through hospital discharge up to 3 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 2 | 0
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.50, Chi-squared

13. Secondary Outcome: Birth Weight
Description: Weight in grams at delivery
Time Frame: Delivery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
grams | 2637 (480) | 2654 (484)
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Birth Weight Less Than 10th Percentile
Description: Neonates whose birth weight is less than the 10th percentile at delivery
Time Frame: Delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 255 | 220
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.13, Chi-squared; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.96 to 1.34]

15. Secondary Outcome: Gestational Age at Delivery
Description: Number of neonates delivered at ≤ 34 weeks 6 days, between 35 weeks 0 days and 35 weeks 6 days, between 36 weeks 0 days and 36 weeks 6 days, between 37 weeks 0 days and 38 weeks 6 days, or on or after 39 weeks 0 days
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants
  ≤34 weeks 6 days | 193 | 213
  35 weeks 0 days to 35 weeks 6 days | 394 | 386
  36 weeks 0 days to 36 weeks 6 days | 609 | 568
  37 weeks 0 days to 38 weeks 6 days | 202 | 185
  ≥39 weeks 0 days | 29 | 48
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.10, Chi-squared

16. Secondary Outcome: Number of Neonates With Necrotizing Enterocolitic (NEC)
Description: Defined as modified Bell Stage 2 or 3. Stage 2: Clinical signs and symptoms with pneumatosis intestinalis on radiographs. Stage 3: Advanced clinical signs and symptoms, pneumatosis, impending or proven intestinal perforation.
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 0 | 1

17. Secondary Outcome: Number of Infants With Neonatal Sepsis
Description: Clinical suspicion of systemic infection with a positive blood, cerebral spinal fluid, or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evience of cardiovascular collapse or an X-ray confirming infection.
Time Frame: Delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 9 | 11
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.62, Chi-squared; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.33 to 1.93]

18. Secondary Outcome: Number of Neonates With Intraventricular Hemorrhage
Description: Grade 3 or 4 Intraventricular Hemorrhage
Time Frame: Delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 2 | 0

19. Secondary Outcome: Neonatal Morbidity Composite
Description: A composite endpoint of morbidities known to be affected by steroid administration will also be evaluated. Specifically, this composite will include RDS, intraventricular hemorrhage (IVH), and NEC
Time Frame: Delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 81 | 90
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.40, Chi-squared; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.66 to 1.18]

20. Secondary Outcome: Number of Neonates With Hypoglycemia
Description: Glucose < 40 mg per deciliter (2.2 mmol per liter) at any time
Time Frame: Delivery through hospital discharge up to 3 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 343 | 210
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Ratio (RR) = 1.60, 95% CI 2-sided [1.37 to 1.87]

21. Secondary Outcome: Time Until First Neonatal Feeding
Description: Median length of time from delivery until the first neonatal feeding
Time Frame: Delivery to 36 hours post delivery
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
hours | 5.5 [1.4 to 24.7] | 9.9 [1.7 to 29.1]
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Neonatal Feeding Difficulty
Description: Inability of the neonate to take all feeds (po), i.e. requiring gavage feeds or IV supplementation.
Time Frame: Delivery to 36 hours post delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 211 | 223
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.40, Chi-squared; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.78 to 1.10]

23. Secondary Outcome: Neonatal Hyperbilirubinemia
Description: Peak total bilirubin of at least 15 mg% or the use of phototherapy.
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 167 | 140
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.15, Chi-squared; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.95 to 1.40]

24. Secondary Outcome: Number of Neonates With Hypothermia
Description: Rectal temperature < 36 C at any time
Time Frame: Delivery through discharge up to 3 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants | 132 | 112
Statistical Analysis 1: Comparison: Betamethasone; Test type: Superiority or Other; p = 0.24, Chi-squared; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.91 to 1.47]

25. Secondary Outcome: Length of NICU or Nursery Stay
Description: Includes need for NICU or intermediate care admission and length of stay if admitted. For analysis purposes, death before discharge is assigned maximum rank
Time Frame: Delivery through hospital discharge up to 3 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants
  NICU stay of any duration | 596 | 629
  NICU stay of ≥3 days | 470 | 518
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Analysis for NICU stay of any duration; Test type: Superiority or Other; p = 0.09, Chi-squared; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.85 to 1.01]
Statistical Analysis 2: Comparison: Betamethasone vs Placebo; Analysis for duration greater than or equal to 3 days; Test type: Superiority or Other; p = 0.03, Chi-squared; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.80 to 0.98]

26. Secondary Outcome: Median Length of Hospital Stay
Description: Median length of maternal hospital stay following delivery
Time Frame: Duration of hospital stay following delivery up to 2 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
days | 7 [4 to 12] | 8 [4 to 13]
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Maternal Outcomes (Participant-based)
Description: Chorioamnionitis: clinical diagnosis and a body temperature of at least 100.4 degrees F., Endometritis: persistent postpartum temperature greater than 100.4 degrees F with uterine tenderness, cesarean delivery
Time Frame: Labor and delivery through 72 hours post partum
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Participants
  Chorioamnionitis | 20 | 32
  Postpartum Endometritis | 16 | 16
  Cesarean Delivery | 454 | 431
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Statistical analysis for chorioamnionitis; Test type: Superiority or Other; p = 0.08, Chi-squared; Risk Ratio (RR) = 0.61, 95% CI 2-sided [0.35 to 1.07]
Statistical Analysis 2: Comparison: Betamethasone vs Placebo; Analysis for Postpartum Endometritis; Test type: Superiority or Other; p = 0.96, Chi-squared; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.49 to 1.95]
Statistical Analysis 3: Comparison: Betamethasone vs Placebo; Statistical analysis for cesarean delivery; Test type: Superiority or Other; p = 0.56, Chi-squared; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.93 to 1.15]

28. Secondary Outcome: Hours From Randomization to Delivery
Description: Median interval of hours from randomization to delivery
Time Frame: Randomization through delivery
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
Hours | 33.0 [15.2 to 111.6] | 30.6 [14.6 to 111.0]
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Analysis for interval from randomization to delivery; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Median Length of Maternal Hospital Stay
Description: Median length of maternal hospital stay in days
Time Frame: Delivery through hospital discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Betamethasone | Placebo
Number analyzed (Participants) | 1427 | 1400
days | 3 [3 to 5] | 3 [3 to 5]
Statistical Analysis 1: Comparison: Betamethasone vs Placebo; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of randomization into the study through 72 hours after delivery.
Description: Adverse events were documented by research nurse coordinators and principal investigators on standardized study protocol forms and reported to the study sponsor. Non-serious adverse events are reported for patients who received 1 or 2 doses of drug or placebo. Not all participants who were randomized received a study injection.
Arm/Group | Betamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 2/1429 | 0/1402
Serious Adverse Events (participants affected / at risk) | 13/1429 | 12/1402
Other Adverse Events (participants affected / at risk) | 223/1428 | 352/1397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Betamethasone (N=1429) | Placebo (N=1402)
Postpartum Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 7 | 5 — Postpartum Hemorrhage
Hypotension (Vascular disorders) | 0 | 1 — Low blood pressure
Seizure (Pregnancy, puerperium and perinatal conditions) | 1 | 1 — Postpartum pregnancy complication
Uterine rupture (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Pregnancy complication
Delayed pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Pregnancy complication
Aortic dissection type 1 (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 2
Obstructed bowel (Gastrointestinal disorders) | 1 | 0 — Maternal obstructed bowel
Lumbar plexus stretch injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — Maternal stretch injury
Neonatal Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neonatal death (General disorders) | 2 | 0 — Two infants died after 72 hours of life but before hospital discharge.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betamethasone (N=1428) | Placebo (N=1397)
Skin reaction at injecton site (Skin and subcutaneous tissue disorders) | 223 (223) | 352 (352) — Pain, bruising, swelling or other local reaction at the injection site with first and/or second dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less